CLINICAL TRIAL: NCT05617690
Title: Effect of Cyclopol on Intraoperative Electrophysiological Monitoring in Spine Surgery: A Randomized Controlled, Noninferiority Study
Brief Title: Cyclopol on Electrophysiological Monitoring During Spine Surgery: a Randomized Controlled, Noninferiority Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: mjj20221108
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Visual Evoked Potentials
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclopol group (Experimental)
  Interventions: Drug: Cyclopol
- Propofol group (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Cyclopol — Cyclopol 0.4mg/kg, sufentanil 0.2-0.4ug/kg and rocuronium 0.6mg/kg will be used for anesthesia induction. Anesthesia maintenance strategy is cyclopol 0.8-2.4 mg/kg/h and remifentanil 0.15 - 0.2 μg/kg/h
  Arms: Cyclopol group
Drug: Propofol — Propofol 1-3mg/kg, sufentanil 0.2-0.4ug/kg and rocuronium 0.6mg/kg will be used for anesthesia induction. The anesthesia maintenance strategy is propofol 4-8mg/kg/h and remifentanil 0.15 - 0.2 μ g/kg/h
  Arms: Propofol group

SUMMARY:
Postoperative visual function injury occurs after spinal cord, neurosurgery, ophthalmology and other operations, which directly affects the postoperative quality of life of patients. Flash visual evoked potential (FVEP) is important for evaluating visual function under general anesthesia during operation. The changes of visual function can be observed and recognized in time through the amplitude changes of FVEP, which can avoid or reduce the visual function damage during operation. Anesthesia method determines the success and variability of electrophysiological monitoring to a certain extent. The purpose of this study is to investigate the effect of total intravenous anesthesia based on cyclopol on FVEP compared with propofol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective spinal surgery under general anesthesia;
2. Intraoperative electrophysiological monitoring is required;
3. 18-65 years old;
4. ASA I-III;
5. Sign the informed consent.

Exclusion Criteria:

1. Patients with visual impairment;
2. Patients with severe liver or kidney disease;
3. Uncontrolled hypertension, diabetes, severe arrhythmia or unstable angina pectoris;
4. Have mental illness or unable to communicate;
5. BMI≥30kg/㎡;
6. Abuse of analgesics and drug abuse history;
7. Muscle weakness, motor dysfunction or neuromuscular junction disease before operation;
8. Preoperative somatosensory dysfunction;
9. Retain trachea catheter after operation;
10. Narcotic drugs and silicone allergy;
11. Visual evoked potential monitoring was rejected.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
N75-p100 amplitude of FVEP | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China